CLINICAL TRIAL: NCT04293068
Title: Effect of Reproductive Tract Microbiota on Pregnancy Outcome in Patients Accepted In-vitro Fertilization/Intracytoplasmic Sperm Injection and Embryo Transfer
Brief Title: Effect of Reproductive Tract Microbiota on Pregnancy Outcome in IVF/ICSI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Li Rong, Director of Reproductive Medical Center, Peking University Third Hospital
Other Study IDs: 2020Microbiota
Record Dates: First submitted 2020-02-27; First posted 2020-03-03 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Infertility; Recurrent Implantation Failure; Recurrent Miscarriage
Keywords: Infertility; Recurrent implantation failure; Recurrent spontaneous abortion; Reproductive tract microbiota; In vitro fertilization
MeSH Terms: conditions — Infertility; Abortion, Habitual; Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Control group: Related tests were normal, because the male factor alone required the first IVF/ICSI cycle; Follow-up of included patients was conducted to determine whether embryo transplantation was performed, and the score of transferred embryos was recorded, and the final control group would be confirmed after achieving clinical pregnancy
- Recurrent implantation failure: Previous ≥3 consecutive embryo transfer failures
- Recurrent spontaneous abortion(miscarriage): ≥2 consecutive spontaneous abortions or embryo damage

SUMMARY:
A single center，observational cohort study to explore the relationship between reproductive tract microbiota and pregnancy outcome in the patients accepted IVF/ICSI. To investigate whether there is a correlation between reproductive tract microbiota and IVF/ICSI outcomes. Whether there are differences in reproductive tract microbiota (such as vagina, follicular fluid, uterine cavity, etc.) in patients with different pregnancy outcomes.

DETAILED DESCRIPTION:
A single center，observational cohort study will enroll 120 infertile participants and then divide them into 3 groups: 1)Male infertility；2)Recurrent implantation failure; 3)Recurrent spontaneous abortion. The study will last for 1 year and recruit participants in Reproductive medicine center of Peking university third hospital. Each participant will be followed up for at least 1 year. Collect samples and record information at the first month, then follow-up 2 months to record the pregnancy outcomes. DNA will be extracted from the samples and then have sequence to figure out the compositions of microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. The sampling cycle of all samples requires no use of glucocorticoids, antibiotics and vaginal drugs within the cycle of this month; No cervical treatment within a week; No irrigation, asexual life within 5 days; Strict contraception in this month;
2. Male infertility (Related tests were normal, because the male factor alone required the first IVF/ICSI cycle; Follow-up of included patients was conducted to determine whether embryo transplantation was performed, and the score of transferred embryos was recorded, and the final control group would be confirmed after achieving clinical pregnancy) OR Recurrent implantation failure (Previous ≥3 consecutive embryo transfer failures) OR Recurrent spontaneous abortion (≥2 consecutive spontaneous abortions or embryo damage)

Exclusion Criteria:

1. Acute genital tract inflammation (including vagina, cervix, endometrium and pelvic cavity)
2. Previous diagnosis of intrauterine adhesion or mechanical damage to the endometrium; drugs and surgery can not restore the function (endometrium thickness <7mm in the window period before transplantation)
3. Untreated hydrosalpinx, submucosal or >4cm intramuscular uterine fibroids, adenomyosis, stage III-IV endometriosis confirmed by surgery, endometritis diagnosed by pathology and other definite factors might affect implantation
4. Chromosomal abnormalities in couples may lead to miscarriage, fetal malformation and other diseases
5. Previous examination indicated the existence of DOR (FSH≥9U/L and/or AMH ≤1.1ng/ml and/or AFC≤5-7)
6. Those with polycystic ovary syndrome, high prolactinemia and other ovulation disorders
7. Those with congenital adrenal hyperplasia, hypothyroidism/hyperthyroidism, diabetes, metabolic syndrome and other endocrine and metabolic diseases
8. BMI less than 18 or more than 25
9. Previous autoimmune diseases such as anti-heart coagulation syndrome, sjogren's syndrome and rheumatoid arthritis
10. Prethrombotic hypercoagulability or family history of thrombosis
11. Female genital tract deformities (whether or not surgically corrected)
12. Those within the programme of oocyte or sperm donor
13. Those with previous history of various types of cancer or serious systemic diseases (such as heart, lung and blood diseases) or mental diseases

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: The recruited participants conformed to the eligibility criteria will be divided into 3 groups (Control group: male infertility; RIF group; RM group). Each group will be recruited at least 30 cases.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 4 weeks after embryo transfer
  One or more observed gestational sac or definitive clinical signs of pregnancy under ultrasonography at 4 weeks after embryo transfer (including clinically documented ectopic pregnancy)

SECONDARY OUTCOMES:
Microbiota ratio | About 2 months later after samples collection
  The ratio of microbiota within 3 groups will be acquired and analyzed by Metagenomics and 16SrRNA sequence. Shannon's diversity index and Chao richness will be used to measure the different ratio of microbiota within these 3 groups
Oocyte retrieval | 36 hours after HCG injection
  Number of oocytes retrieved for use in the following IVF-ET procedure will be counted under microscope
Fertilization rate | 16-20 hours after oocyte retrieval
  Number of zygotes with 2 PN will be observed and counted under microscope
Available embryo | 72 hours after oocyte retrieval
  Number of embryos ≥4 cells and ≤30% fragmentation on day 3 observation will be observed and counted under microscope
Good quality embryo | 72 hours after oocyte retrieval
  Number of embryos with ≥6 cells and ≤30% fragmentation developed from 2PN embryos on day 3 observation
Endometrium thickness | On the day of embryo transfer
  Transvaginal Ultrasonography will be used to measure the endometrium thickness on the day of embryo transfer
Implantation rate | 30 days after embryo transfer
  Number of gestational sacs observed per embryo transferred will be observed under ultrasonography
Ongoing pregnancy rate | 10 weeks after embryo transfer
  Presence of a gestational sac and fetal heartbeat after 10 weeks of gestationwill be monitored by ultrasound
Live birth rate | After 24 weeks of gestation
  A delivery of one or more living infants (≥24 weeks gestation or birth weight more than 1,000g) will be followed up via telephone

CONTACTS AND LOCATIONS:
Overall Officials: Rong Li, M.D., Study Director — Peking University Third Hospital
Locations (1):
- Peking university third hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided